CLINICAL TRIAL: NCT00162955
Title: The Multi-centers Trial for Patients With Non-Hodgkin's Lymphoma to Assess the Protective Effect of Valsartan on Chronic Cardiotoxicity Induced by CHOP
Brief Title: Prevention of CHOP-induced Chronic Cardiotoxicity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Osaka City University (Other)
Responsible Party: Hirohisa Nakamae, MD. PhD., Osaka City University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OLSG-0401
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2010-09

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: untreated adult Non-Hodgkin's Lymphoma; CHOP protocol; Angiotensin II Type 1 Receptor Blockers; Cardiomyopathy
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Cardiomyopathies | interventions — Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARB administration (Experimental): 80mg/day from the day of the start of 1st CHOP until the completion of all the evaluations
  Interventions: Drug: Valsartan
- non-administration (No Intervention): ARB non-administration group

INTERVENTIONS:
Drug: Valsartan — Patients allocated into ARB administration group take Valsartan (80mg/day) from the day of the start of 1st CHOP until the completion of all the evaluations.
  Other Names: Diovan
  Arms: ARB administration

SUMMARY:
The purpose of this study is to assess the protective effect of Valsartan on chronic cardiotoxicity induced by CHOP.

DETAILED DESCRIPTION:
Doxorubicin has been one of the most important key drugs in treatment for malignancies. However, its use is limited by dose-dependent cumulative cardiotoxicity. This multi-centers trial was designed to investigate the preventive effect of Valsartan, the angiotensin II type 1 receptor blocker (ARB) on chronic cardiotoxicity due to doxorubicin based chemotherapy. Patients with untreated non-Hodgkin's lymphoma who are scheduled to receive at least 6 courses of the standard CHOP (-R) will be randomized by the minimization methods to the treatment group with Valsartan (80mg once daily by oral during entire 6 courses of CHOP) or control group. Cardiac function will be evaluated in detail before and after 3 and 6 courses of CHOP (-R).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of non-Hodgkin's lymphoma (NHL)
* Untreated lymphoma
* Performance status from 0 to 1,
* Total serum bilirubin < 2.0 mg/dl
* Serum creatinine level < 2.0 mg/dl
* Ejection fraction of the left ventricle >50 %
* Systolic blood pressure at rest being 90 mmHg or more

Exclusion Criteria:

* Severe complication including chronic or acute heart failure, angina, old myocardial infarction, liver cirrhosis, and interstitial pneumonia
* Pregnancy, nursing mothers or women of child-bearing potential
* Hypertension under medication
* Diabetes mellitus under medication
* Hyperthyroidism, nephrotic syndrome, Cushing's syndrome
* Atrial arrythmias
* Severe psychopathy
* Cerebrovascular accidents within the past 3 months
* Positive serum HBs antigen or HCV antibody
* A history of renal failure
* A contraindication to A-II antagonists or noncompliance
* Treatment with any of the following drugs within the past 3 months : A-II antagonists, ACE inhibitors, vitamin E, probucol, calcium antagonists, beta-blockers, and steroid pulse therapy.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2004-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Cardiac Event after 3rd and 6th course of CHOP(-R) | Basically 14-21 (at a maximum 28) days after the start of 3rd and 6th course of CHOP(-R).

SECONDARY OUTCOMES:
Changes of ECG, UCG and serum markers after 3 and 6 courses of CHOP (-R) | 14-21 (at a maximum 28) days after the start of 3rd and 6th course of CHOP(-R).

CONTACTS AND LOCATIONS:
Overall Officials: Masayuki Hino, MD, PhD, Study Chair — Graduate School of Medicine, Osaka City University; Hirohisa Nakamae, MD, PhD, Principal Investigator — Graduate School of Medicine, Osaka City University
Locations (1):
- Graduate School of Medicine, Osaka City University, Osaka, Osaka, Japan

REFERENCES:
- [Background] Toko H, Oka T, Zou Y, Sakamoto M, Mizukami M, Sano M, Yamamoto R, Sugaya T, Komuro I. Angiotensin II type 1a receptor mediates doxorubicin-induced cardiomyopathy. Hypertens Res. 2002 Jul;25(4):597-603. doi: 10.1291/hypres.25.597. PMID 12358147